CLINICAL TRIAL: NCT03286946
Title: The Difference of Intravascular Injection Rate During Cervical Transforaminal Epidural Block Using Blunt-type Block Needle Compared to Sharp-type Block Needle.
Brief Title: Detection of Intravascular Injection Between Blunt and Sharp Needles During Cervical Transforaminal Epidural Block.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Saeyoung Kim, MD, PhD, Associate professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2016-09-009
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Pain; Radicular; Neuropathic, Cervical
MeSH Terms: conditions — Pain | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blunt-type block needle (Experimental): block with Blunt-type block needle.
  Interventions: Procedure: block with Blunt-type block needle.
- Sharp-type block needle (Active Comparator): block with Sharp-type block needle.
  Interventions: Procedure: block with sharp-type block needle.

INTERVENTIONS:
Procedure: block with Blunt-type block needle. — Under fluoroscopic guidance, cervical transforaminal epidural injections were performed using 22 gauge blunt needle. The needle position was confirmed using biplanar fluoroscopy and 2 ml of nonionic contrast media was injected to detect intravascular injection.
  Arms: Blunt-type block needle
Procedure: block with sharp-type block needle. — Under fluoroscopic guidance, cervical transforaminal epidural injections were performed using 22 gauge sharp needle. The needle position was confirmed using biplanar fluoroscopy and 2 ml of nonionic contrast media was injected to detect intravascular injection.
  Arms: Sharp-type block needle

SUMMARY:
This study evaluates the incidence of intravascular injection during cervical transforaminal epidural block using blunt needle, compared to the sharp needle. The investigators will performed cervical transforaminal epidural block using blunt-type block needle in half of participants or sharp-type block needle in the other half.

DETAILED DESCRIPTION:
Cervical transforaminal epidural block is an effective treatment option of radiating pain. There are potential risks associated with transforaminal epidural block such as infection, dural puncture, bleeding, and intravascular injection. Although the risk is low, intravascular injection should be carefully monitored because intravascular injection of particulate steroids can cause fatal neurologic deficits such as spinal infarction and cerebral infarction.

The incidence of intravascular injection during transforaminal epidural block with real time fluoroscopy guidance depends on spinal level. The previous studies using real time fluoroscopy demonstrated that the incidence of intravascular injection of cervical transforaminal epidural block is higher than that of lumbosacral transforaminal epidural block.

In this study, therefore, the investigators investigate the incidence of intravascular injection during cervical transforaminal epidural block using blunt needle, compared to the sharp needle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiating pain from cervical spinal stenosis and herniated nucleus pulposus.

Exclusion Criteria:

* Pregnancy, allergic to contrast media, patient refusal, and patients with persistent contraindication to nerve block such as coagulopathy and infection of the injection site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Intravascular injection | During procedure
  Intravascular injection was defined as contrast media spreading out through the vascular channel during injection of contrast media under real time fluoroscopy. The investigators observed the intravascular injection during the procedure. The intravascular injection rate was calculated based on the total number of treated levels.

SECONDARY OUTCOMES:
Needling time | During procedure
  Needling time for both the sharp and blunt needles was started upon insertion of the needle through the skin and ended upon injection of contrast media under real time fluoroscopy.